CLINICAL TRIAL: NCT04131218
Title: Pharmacokinetics and Pharmacodynamics of Sugammadex in Reversal of Vecuronium-induced Neuromuscular Blockade in Anesthesia Obese Patients Undergoing Bariatric Surgery
Brief Title: Pharmacokinetics and Pharmacodynamics of Sugammadex in Reversal of Vecuronium-induced Neuromuscular Blockade
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, Clinical Professor, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PK and PD of Sug
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pharmacokinetics; Pharmacodynamics
Keywords: Sugammadex; Obese
MeSH Terms: conditions — Obesity | interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Obese group (Experimental): n=8, 25≤BMI≤39.9kg/m²
  Interventions: Drug: Sugammadex
- Morbidly obese group (Experimental): n=8, BMI≥40kg/m²
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — Each patient received a single dose administration of sugammadex 2mg/kg according to the ideal body weight (IBW) at reappearance of the second twitch of the train-of-four (TOF).
  Other Names: Bridion; Org 25969

SUMMARY:
The purpose of this study is to illustrate pharmacokinetics and pharmacodynamics of sugammadex in reversal of vecuronium-induced neuromuscular blockade in anesthesia obese patients undergoing bariatric surgery.

DETAILED DESCRIPTION:
16 obese patients undergoing bariatric surgery were divided into 2 groups according to body mass index (BMI), including obese group (O group, n=8, 25≤BMI≤39.9kg/m²) and morbidly obese group (M group, n=8, BMI≥40kg/m²).

Vecuronium was continuous infusing to maintain moderate neuromuscular blockade during the laparoscopic surgery and stopped infusing after the laparoscopic procedure. A single dose administration of sugammadex (Sug) 2.0mg/kg according to ideal body weight (IBW) was given at the reappearance of the second twitch of the train-of-four (TOF) response.

On one hand, venous blood samples were obtained before administration of Sug and at 2, 3, 5, 10, 15, 20, 30, 60 minutes and 2, 4, 6, 8 hours after administration of Sug to determine plasma concentration of Sug using HPLC-MS. On the other hand, time from start of administration of Sug to recovery of TOF ratio to 0.9 and other clinical indicators were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA: Ⅰ~Ⅲ
* BMI≥25kg/m²
* Patients receiving bariatric surgery.

Exclusion Criteria:

* Pregnant or lactating women
* Neuromuscular diseases
* Malignant hyperthermia or allergic history during general anesthesia
* Drugs that react with rocuronium and vecuronium were taken

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of Sugammadex | 0, 2, 3, 5, 10, 15, 20, 30, 60 minutes and 2, 4, 6, 8 hours
  venous blood samples were obtained
Recovery Time and TOF ratio | TOF ratio at 30, 60, 90, 120, 150 seconds after administration
  time from start of administration of Sug to recovery of TOF ratio to 0.9 and other indicators

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Background] GBD 2015 Obesity Collaborators; Afshin A, Forouzanfar MH, Reitsma MB, Sur P, Estep K, Lee A, Marczak L, Mokdad AH, Moradi-Lakeh M, Naghavi M, Salama JS, Vos T, Abate KH, Abbafati C, Ahmed MB, Al-Aly Z, Alkerwi A, Al-Raddadi R, Amare AT, Amberbir A, Amegah AK, Amini E, Amrock SM, Anjana RM, Arnlov J, Asayesh H, Banerjee A, Barac A, Baye E, Bennett DA, Beyene AS, Biadgilign S, Biryukov S, Bjertness E, Boneya DJ, Campos-Nonato I, Carrero JJ, Cecilio P, Cercy K, Ciobanu LG, Cornaby L, Damtew SA, Dandona L, Dandona R, Dharmaratne SD, Duncan BB, Eshrati B, Esteghamati A, Feigin VL, Fernandes JC, Furst T, Gebrehiwot TT, Gold A, Gona PN, Goto A, Habtewold TD, Hadush KT, Hafezi-Nejad N, Hay SI, Horino M, Islami F, Kamal R, Kasaeian A, Katikireddi SV, Kengne AP, Kesavachandran CN, Khader YS, Khang YH, Khubchandani J, Kim D, Kim YJ, Kinfu Y, Kosen S, Ku T, Defo BK, Kumar GA, Larson HJ, Leinsalu M, Liang X, Lim SS, Liu P, Lopez AD, Lozano R, Majeed A, Malekzadeh R, Malta DC, Mazidi M, McAlinden C, McGarvey ST, Mengistu DT, Mensah GA, Mensink GBM, Mezgebe HB, Mirrakhimov EM, Mueller UO, Noubiap JJ, Obermeyer CM, Ogbo FA, Owolabi MO, Patton GC, Pourmalek F, Qorbani M, Rafay A, Rai RK, Ranabhat CL, Reinig N, Safiri S, Salomon JA, Sanabria JR, Santos IS, Sartorius B, Sawhney M, Schmidhuber J, Schutte AE, Schmidt MI, Sepanlou SG, Shamsizadeh M, Sheikhbahaei S, Shin MJ, Shiri R, Shiue I, Roba HS, Silva DAS, Silverberg JI, Singh JA, Stranges S, Swaminathan S, Tabares-Seisdedos R, Tadese F, Tedla BA, Tegegne BS, Terkawi AS, Thakur JS, Tonelli M, Topor-Madry R, Tyrovolas S, Ukwaja KN, Uthman OA, Vaezghasemi M, Vasankari T, Vlassov VV, Vollset SE, Weiderpass E, Werdecker A, Wesana J, Westerman R, Yano Y, Yonemoto N, Yonga G, Zaidi Z, Zenebe ZM, Zipkin B, Murray CJL. Health Effects of Overweight and Obesity in 195 Countries over 25 Years. N Engl J Med. 2017 Jul 6;377(1):13-27. doi: 10.1056/NEJMoa1614362. Epub 2017 Jun 12. PMID 28604169
- [Background] Hanley MJ, Abernethy DR, Greenblatt DJ. Effect of obesity on the pharmacokinetics of drugs in humans. Clin Pharmacokinet. 2010;49(2):71-87. doi: 10.2165/11318100-000000000-00000. PMID 20067334
- [Background] Suy K, Morias K, Cammu G, Hans P, van Duijnhoven WG, Heeringa M, Demeyer I. Effective reversal of moderate rocuronium- or vecuronium-induced neuromuscular block with sugammadex, a selective relaxant binding agent. Anesthesiology. 2007 Feb;106(2):283-8. doi: 10.1097/00000542-200702000-00016. PMID 17264722
- [Background] Sanfilippo M, Alessandri F, Wefki Abdelgawwad Shousha AA, Sabba A, Cutolo A. Sugammadex and ideal body weight in bariatric surgery. Anesthesiol Res Pract. 2013;2013:389782. doi: 10.1155/2013/389782. Epub 2013 Jun 6. PMID 23840203
- [Background] Asztalos L, Szabo-Maak Z, Gajdos A, Nemes R, Pongracz A, Lengyel S, Fulesdi B, Tassonyi E. Reversal of Vecuronium-induced Neuromuscular Blockade with Low-dose Sugammadex at Train-of-four Count of Four: A Randomized Controlled Trial. Anesthesiology. 2017 Sep;127(3):441-449. doi: 10.1097/ALN.0000000000001744. PMID 28640017
- [Background] Staals LM, Snoeck MM, Driessen JJ, van Hamersvelt HW, Flockton EA, van den Heuvel MW, Hunter JM. Reduced clearance of rocuronium and sugammadex in patients with severe to end-stage renal failure: a pharmacokinetic study. Br J Anaesth. 2010 Jan;104(1):31-9. doi: 10.1093/bja/aep340. PMID 20007792